CLINICAL TRIAL: NCT00182104
Title: An International Multi Centre Randomized Clinical Trial Of Anticoagulation In Children Following Fontan Procedures
Brief Title: International Multi Centre Randomized Clinical Trial Of Anticoagulation In Children Following Fontan Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CTMG-1998-Fontan; Hearth and Stroke grant 1998
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Heart Defect; Triscupid Atresia
Keywords: Fontan procedure; Anticoagulation; Thrombosis; Thromboembolism; Prevention
MeSH Terms: conditions — Thrombosis; Thromboembolism

INTERVENTIONS:
Drug: Warfarin vs ASA

SUMMARY:
Compare heparin/warfarin to ASA for thromboembolic prophylaxis in the first two years following Fontan procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is scheduled to have a Fontan or modified Fontan procedure

Exclusion Criteria:

1. Requirement for long-term anticoagulation (e.g., prosthetic heart valve, active DVT)
2. Risk of significant bleeding or any other known medical contraindication to Heparin, Warfarin, or ASA.
3. Inability to supervise therapy due to social or geographical reasons.
4. Pregnancy or potential pregnancy during study period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 111
Dates: Start 1998-08; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Warfarin vs ASA in prevention of thrombosis 2 yrs after Fontan

SECONDARY OUTCOMES:
Identify subpopulation of Fontan pts at high risk for TEs
Determine high risk period for TEs in first 2 yrs post Fontan

CONTACTS AND LOCATIONS:
Overall Officials: Paul Monagle, MD, Study Chair — Royal Children's Hospital, Parkville, Victoria, Australia; Brian McCrindle, MD, Principal Investigator — The Hospital for Sick Children; Robin Roberts, MD, Principal Investigator — McMaster University
Locations (7):
- Royal Children's Hospital, Parkville, Victoria, Australia
- Canada (6):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta HSC, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - Sick Children's Hospital, Toronto, Ontario
  - Hopital Ste-Justine, Montreal, Quebec

REFERENCES:
- [Derived] McCrindle BW, Manlhiot C, Cochrane A, Roberts R, Hughes M, Szechtman B, Weintraub R, Andrew M, Monagle P; Fontan Anticoagulation Study Group. Factors associated with thrombotic complications after the Fontan procedure: a secondary analysis of a multicenter, randomized trial of primary thromboprophylaxis for 2 years after the Fontan procedure. J Am Coll Cardiol. 2013 Jan 22;61(3):346-53. doi: 10.1016/j.jacc.2012.08.1023. Epub 2012 Dec 12. PMID 23246393
- [Derived] Monagle P, Cochrane A, Roberts R, Manlhiot C, Weintraub R, Szechtman B, Hughes M, Andrew M, McCrindle BW; Fontan Anticoagulation Study Group. A multicenter, randomized trial comparing heparin/warfarin and acetylsalicylic acid as primary thromboprophylaxis for 2 years after the Fontan procedure in children. J Am Coll Cardiol. 2011 Aug 2;58(6):645-51. doi: 10.1016/j.jacc.2011.01.061. PMID 21798429